CLINICAL TRIAL: NCT05670379
Title: A Randomized, Parallel-Group Study to Assess the Safety, Tolerability, and Pharmacokinetics of Exenatide Implant
Brief Title: Assessment of Safety, Tolerability and Drug Levels of Exenatide Implant
Acronym: LIBERATE-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vivani Medical, Inc (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VANI-NP-001
Record Dates: First submitted 2022-12-13; First posted 2023-01-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Overweight and Obesity; Type2diabetes
MeSH Terms: conditions — Overweight; Obesity | interventions — Exenatide; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Exenatide Implant (Experimental): One Exenatide Implant that delivers approximately 52 microgram/day of exenatide will be inserted subdermally just under the skin of the upper outer arm for the 9-week treatment period.
  Interventions: Combination Product: Exenatide Implant
- Bydureon BCise (exenatide extended release) (Active Comparator): 2 mg subcutaneous injection every week for a duration of 9 weeks
  Interventions: Drug: Bydureon BCise (exenatide extended release)
- Semaglutide (Active Comparator): 1.0 mg subcutaneous injection every week for a duration of 9 weeks
  Interventions: Drug: Semaglutide, 1.0 mg/mL

INTERVENTIONS:
Combination Product: Exenatide Implant — Exenatide Implant is a drug:device combination that delivers steady levels of exenatide, a glucagon-like peptide-1(GLP-1) receptor agonist, for an extended period of time following subdermal insertion.
  Other Names: NPM115/NPM119
  Arms: Exenatide Implant
Drug: Bydureon BCise (exenatide extended release) — glucagon-like peptide-1 (GLP-1) receptor agonist
  Arms: Bydureon BCise (exenatide extended release)
Drug: Semaglutide, 1.0 mg/mL — glucagon-like peptide-1 (GLP-1) receptor agonist
  Other Names: Wegovy, Ozempic
  Arms: Semaglutide

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and drug levels of an exenatide implant administered subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27 to 40 kg/m^2
* Estimated glomerular filtration rate (eGFR) >/= 90 mL/min/1.73 m^2
* HbA1c < 6.0% and FPG < 6.7 mol/L

Exclusion Criteria:

* Has a clinically significant medical condition that could potentially affect study participation and/or personal well-being
* History of Type 1 or Type 2 Diabetes
* History of, or currently has, acute or chronic pancreatitis or has triglyceride concentrations ≥500 mg/dL
* Has medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia (MEN II) or a family history of MTC or MEN II
* Current or past exposure to exenatide

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | 9 weeks
  Total exenatide concentration
Maximum plasma concentration observed (Cmax) | 9 weeks
  Maximal exenatide concentration
Time to maximum plasma concentration observed (Tmax) | 9 weeks
  Time to reach maximal exenatide concentration
Adverse events | 9 weeks
  Incidence of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Vivani Medical, Inc
Locations (1):
- CMax, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No